CLINICAL TRIAL: NCT05355480
Title: Advanced Machine Learning Analysis of Handwriting in Patients With Movement Disorders
Brief Title: Handwriting Analysis in Movement Disorders
Acronym: HANDWRML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Suppa, Prof., Neuromed IRCCS
Other Study IDs: NEUR_04
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Movement Disorders; Parkinson Disease; Writing Disorder
MeSH Terms: conditions — Movement Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: Collection of handwriting samples
- Patients with Parkinson's disease: Collection of handwriting samples

SUMMARY:
Handwriting is a complex cognitive prowess that deteriorates in patients affected by neurodegenerative diseases, including movement disorders. More in detail, patients with Parkinson's disease (PD) may manifest prominent handwriting abnormalities which have been collectively identified as parkinsonian micrographia. MIcrographia may manifest at the onset of the disease and then worsens progressively with time. Previous techniques released to investigate micrographia in PD relied on perceptual analysis of simple tasks or were based on expensive technological tools, including tablets. However, handwriting can be promptly collected in an ecological scenario, through safe, cheap, and largely available tools. Also, the objective handwriting analysis through artificial intelligence would represent an innovative strategy even superior to previous techniques, since it allows for the analysis of large amounts of data. In this experimental project, the investigators apply a specific machine learning algorithm to analyze handwriting samples recorded in healthy controls and PD patients. The study aims to verify whether the technique proposed by the investigators would be able to detect parkinsonian micrographia objectively, monitor the evolution of handwriting abnormalities and assess the symptomatic improvement of handwriting following L-Dopa administration in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy conditions
* clinical diagnosis of Parkinson's disease

Exclusion Criteria:

* cognitive decline

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and patients with idiopathic PD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke size of handwriting characters | through study completion, an average of 1 year
  height of single letters

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy